CLINICAL TRIAL: NCT02610036
Title: Pilot Study on the Presence of Microangiopathy in Diabetic Foot Ulcer
Brief Title: Obliterating Diabetic Microangiopathy of the Diabetic Foot
Status: Completed | Type: Observational
Sponsor: IRCCS Multimedica (Other)
Responsible Party: Sponsor
Other Study IDs: PROT 18 /2011Cardiovascular
Record Dates: First submitted 2012-03-30; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2012-03

CONDITIONS: Diabetic Foot
Keywords: diabetes; foot ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- neuropathic type 2 diabetic patients: the foot ulcer of 30 neuropathic and 30 neuroischemic type 2 diabetic patients
- neuroischemic type 2 diabetic patients: the foot ulcer of 30 neuropathic and 30 neuroischemic type 2 diabetic patients

SUMMARY:
The purpose of this study will be the assessment of microangiopathy determined by the increase of capillary basement membrane thickness and decrease of capillary lumen area in the foot ulcer of 30 neuropathic and 30 neuroischemic type 2 diabetic patients

DETAILED DESCRIPTION:
Primary endpoint of the study is to quantitatively evaluate the presence of microangiopathy as increase of capillary basement membrane thickness and decrease of capillary lumen area determined by transmission electron microscopy analysis in type 2 diabetic patients with only motor-sensory neuropathy or chronic critical ischemia affected by foot ulcer.

The following parameters will be evaluated:

* presence of capillary (n/mm2) and thrombosis (%) and correlation of this quantitative histological data with ischemic parameters (TcPO2, ankle-brachial index) and risk of diastasis
* correlation between presence of inflammatory infiltrate (leukocytes/mm2) with blood inflammatory parameters (erythrocyte sedimentation rate (ESR), C-reactive protein, alpha-2 globulin)
* rate of diastasis and/or time required for recovery associated with histopathological data
* presence of acanthosis related to clinical and demographic variables

ELIGIBILITY:
Inclusion Criteria:-

* adult type 2 diabetic patients of either gender
* diabetes for more than 10 years
* motor-sensory diabetic neuropathy with or without chronic critical ischemia
* local residents
* ulcer with surgical therapy indication of removal the 1st ray because of gangrene or osteomyelitis

Exclusion Criteria:

* type 1 diabetic patients
* diabetes for less than 10 years
* renal replacement therapy
* urgent surgical procedure for sepsis
* immunosuppressive therapy
* not local residents

  * Cancer with adverse prognosis in months, or chemotheraputic treatment
  * Ongoing or planned pregnancy
  * Lack of consent to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 diabetic patients with only neuropathy, 30 diabetic patients with critical limb ischemia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
presence of microangiopathy | 24 hours after surgical amputation at the first ray level for treatment of foot ulcer
  presence of microangiopathy as increase of capillary basement membrane thickness and decrease of capillary lumen area by transmission electron microscopy in the skin of type 2 diabetic patients with foot ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Ezio Faglia, MD, Principal Investigator — IRCCS Multimedica
Locations (1):
- Diabetic Foot Center - IRCCS Multimedica,, Sesto San Giovanni, (Milan), Italy, Italy

REFERENCES:
- [Derived] Fiordaliso F, Clerici G, Maggioni S, Caminiti M, Bisighini C, Novelli D, Minnella D, Corbelli A, Morisi R, De Iaco A, Faglia E. Prospective study on microangiopathy in type 2 diabetic foot ulcer. Diabetologia. 2016 Jul;59(7):1542-1548. doi: 10.1007/s00125-016-3961-0. Epub 2016 Apr 28. PMID 27121168